CLINICAL TRIAL: NCT00561288
Title: Effects of Acetaminophen on Hurt Feelings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 20619
Record Dates: First submitted 2007-11-16; First posted 2007-11-20 (Estimated); Last update posted 2008-06-25 (Estimated); Status verified 2008-06

CONDITIONS: Emotional Pain
Keywords: Acetaminophen; Social Psychology; Affect; Interpersonal Rejection
MeSH Terms: interventions — Acetaminophen; Starch

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 2000 mg acetaminophen per day
  Interventions: Drug: acetaminophen
- 2 (Placebo Comparator): 2000 mg cornstarch per day
  Interventions: Other: cornstarch

INTERVENTIONS:
Drug: acetaminophen — 2 x 1000 mg doses per day
  Arms: 1
Other: cornstarch — 2 x 1000 mg cornstarch per day
  Arms: 2

SUMMARY:
The purpose of the study is to investigate whether ingestion of acetaminophen reduces the experience of hurt feelings.

ELIGIBILITY:
Inclusion Criteria:

* University of Toronto undergraduate psychology student

Exclusion Criteria:

* Alcohol consumption (more than 2 drinks per day)
* Intake of enzyme-inducing drugs
* Prolonged fasting/eating disorders/gastroenteritis
* Intake of other over-the-counter or prescription analgesics
* Liver Disorders
* History of abuse treatment

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-11; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Self-reported daily hurt feelings | 21 days

SECONDARY OUTCOMES:
Reports of emotional states other than hurt feelings | 21 days
Evaluations of self-worth | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Geoff MacDonald, Ph.D., Principal Investigator — University of Toronto; Nathan DeWall, Ph.D., Principal Investigator — University of Kentucky
Locations (1):
- University of Toronto, Toronto, Ontario, Canada